CLINICAL TRIAL: NCT00670397
Title: Phase I Trial of Photodynamic Therapy With HPPH (2-1[Hexyloxyethyl]-2-devinylpyropheophorbide-a) for Treatment of Dysplasia, Carcinoma in Situ and Stage I Carcinoma of the Oral Cavity
Brief Title: Photodynamic Therapy Using HPPH in Treating Patients With Recurrent Dysplasia, Carcinoma in Situ, or Stage I Oral Cavity Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: safety issues
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 109307; RPCI-I-109307 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2008-04-30; First posted 2008-05-01 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Head and Neck Cancer
Keywords: stage I squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; stage 0 lip and oral cavity cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Mouth Neoplasms | interventions — 2-(1-hexyloxyethyl)-2-devinyl pyropheophorbide-a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (PDT) (Experimental): Patients undergo PDT comprising HPPH IV over 1 hour on day 1 followed by laser light treatment to the tumor bed on day 2. Treatment may repeat every 8 weeks for up to 3 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: HPPH

INTERVENTIONS:
Drug: HPPH — IV

SUMMARY:
RATIONALE: Photodynamic therapy uses a drug, such as HPPH, that is absorbed by tumor cells. The drug becomes active when it is exposed to light. When the drug is active, tumor cells are killed.

PURPOSE: This phase I trial is studying the side effects and best dose of photodynamic therapy using HPPH in treating patients with recurrent dysplasia, carcinoma in situ, or stage I oral cavity cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the maximum tolerated dose in the oral cavity of photodynamic therapy (PDT) using HPPH and 665 nm light in patients with recurrent dysplasia, carcinoma in situ, or stage I squamous cell carcinoma of the oral cavity.

Secondary

* To determine response of dysplasia, carcinoma in situ, and selected patients with T1 squamous cell carcinoma of the oral cavity using PDT with HPPH and 665 nm light.

OUTLINE: This is a dose-escalation study of laser light dose therapy.

Patients receive HPPH IV over 1 hour on day 1. Approximately 24 hours after receiving HPPH, patients undergo laser light treatment to the tumor bed on day 2. Patients with multicentric or large area confluent disease receive a second course of treatment at least 8 weeks later for lesions untreated at the first treatment session.

After completion of study treatment, patients are followed at 1 week, 1 month, 3 months, and periodically thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Biopsy-confirmed diagnosis of 1 of the following:

  * Mild to severe dysplasia
  * Carcinoma in situ (CIS) of the oral cavity

    * Carcinoma must be less than 3mm thick
  * Stage I (T1) squamous cell carcinoma of the oral cavity
* Recurrent or primary disease
* No T2 or greater squamous cell carcinoma, exophytic CIS, or dysplasia lesions

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Total bilirubin ≤ 2.0 mg/dL
* Creatinine ≤ 2.0 mg/dL
* Alkaline phosphatase ≤ 3 times the upper limit of normal (ULN)
* SGOT ≤ 3 times ULN
* Not pregnant
* Fertile patients must use effective contraception
* No porphyria or hypersensitivity to porphyrin or porphyrin-like compounds

PRIOR CONCURRENT THERAPY:

* Prior therapy of any type allowed
* More than 4 weeks since prior and no concurrent chemotherapy or radiotherapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2010-06; Primary Completion 2011-11 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Evidence of dose limiting Toxicities (DLT) | First four weeks
  Each cohort of 3 patients will be observed for the first 4 weeks to monitor for DLT.
Tumor response | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Arshad, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States